CLINICAL TRIAL: NCT02728271
Title: A Pilot Study of Immuno-ablation With Chemoimmunoradiation Followed by Autologous Hematopoietic Progenitor Cell (HPC) Transplant for Adult Subjects With Churg-Strauss Syndrome
Brief Title: Immuno-ablation With Chemoimmunoradiation and Autologous Stem Cell Transplant for Churg-Strauss Syndrome
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: PI left the institution
Sponsor: Mounzer Agha (Other)
Responsible Party: Sponsor-Investigator, Mounzer Agha, Associate Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-146
Record Dates: First submitted 2016-03-14; First posted 2016-04-05 (Estimated); Last update posted 2017-08-01 (Actual); Status verified 2016-03

CONDITIONS: Churg-Strauss Syndrome
MeSH Terms: conditions — Churg-Strauss Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HPC cell infusion (Experimental): Autologous HPC will be infused within 24 hours of completing the chemotherapy. A total of 5 x 106/kg CD34+ HPC will be infused. The remaining HPC will be stored as back-up, to be used in case of graft failure.
  Interventions: Biological: HPC cell infusion

INTERVENTIONS:
Biological: HPC cell infusion — Administration of total lymphatic irradiation, antithymocyte globulins, and high dose cyclophosphamide, followed by the infusion of autologous stem cells.
  Patients will not receive any cyclosporin A, rituximab, or azathioprine post transplant.

SUMMARY:
Churg-Strauss syndrome is a rare autoimmune inflammatory disease affecting medium- and small-sized blood vessels, causing asthma, abnormalities of the blood, lung diseases, and neuropathy. The main cause of death in these patients is heart attack. Without therapy, the 5-year survival in patients with Churg-Strauss syndrome is 25%. Although with the 5-year survival is increased to 62% with the appropriate therapy, many patients remain refractory to therapy. The long term outcome of these patients remains grim.

The aim of this research study is to determine if suppressing the immune system using a combination of high dose chemotherapy, antibodies, and radiation followed by stem cell transplant will abolish the 'bad' immune system and let the patient's body establish a new immune system that does not attack the blood vessels.

DETAILED DESCRIPTION:
Churg-Strauss syndrome is a rare autoimmune inflammatory disease affecting medium- and small-sized arteries and veins and is closely related to Wegener's granulomatosis. It is also one of the diseases that are associated with antibodies to neutrophils cytoplasmic antigens (ANCAs). Patients with Churg-Strauss syndrome often present with refractory asthma, eosinophilia, pulmonary infiltrates and mononeuritis multiplex.

Corticosteroids remain the first line therapy for these patients and most patients respond to corticosteroid therapy. However, a small proportion of patients need other immunosuppressive agents such as cyclophosphamide, cyclosporine A, Rituximab, and azathioprine. Still a number of these patients remain refractory and extremely dependent on high dose corticosteroids.

The principal cause of mortality in these patients is myocarditis and myocardial infarction due to coronary arteritis. Without therapy, the 5-year survival in patients with Churg-Strauss syndrome is 25%. Although with the 5-year survival is increased to 62% with the appropriate therapy, many patients remain refractory to therapy. The long term outcome of these patients remains grim.

In this study, the investigators hypothesize that the addition of total lymphatic irradiation to the combination of high dose cyclophosphamide and antithymocyte globulins can be given safely to these patients and will not only induce disease remission in patients with refractory Churg-Strauss syndrome, it would also induce sustained and long period of medication-free remission in these patients. Since this combination preparative regimen has never been used previously, the investigators will test this hypothesis in a pilot study.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-60, inclusive
* Subjects carry a diagnosis of Churg-Strauss syndrome, with typical clinical, pathologic, and/or radiological appearances.
* Must have a pulmonologist/immunologist providing the primary care for the Churg-Strauss syndrome and be willing to be evaluated for the Churg-Strauss syndrome who is the co-investigator in the protocol.
* Must be documented to be HIV negative.
* Subjects must be able to give written consent.
* Subjects with abscesses are eligible to enroll once the abscesses or any other significant infection has resolved.
* Subjects must not be pregnant and will undergo a pregnancy test prior to starting the study treatment. The subjects should also be willing to take the appropriate contraception starting at least three months prior to the transplant.
* All eligible subjects will need the approval of the insurance company for the coverage of the study treatment.
* Life expectancy of more than 6 months. ECOG performance status of 0 or 1.
* No evidence of myelodysplastic on peripheral blood smear
* Baseline serum creatinine must be <1.5 mg/dL, left ventricular ejection fraction >55%, adequate pulmonary functions (oxygen saturation at room air of >90%), and AST and ALT not > 2x upper limits of normal, and no history of previous or active malignancy, except for localized cutaneous basal or squamous cell carcinoma in situ of the cervix.
* Evidence for life threatening disease, including FEV1 <50% predicted (on therapy) and/or cardiac involvement (arrhythmias, failure)
* Failure to stabilize in response to prednisone (or equivalent) at doses of <20 mg per day
* Failure of at least 3 other immunosuppressives to stabilize disease, including drugs like cyclophosphamide, rituximab, mepolizumab, azathioprine.

Exclusion Criteria:

* Failure to accept or comprehend irreversible sterility as a potential side effect of therapy.
* Previous allergy to cyclophosphamide, rituximab, mepolizumab, azathioprine.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2016-07-22 (Actual); Study Completion 2016-08-20 (Actual)

PRIMARY OUTCOMES:
number of patients with adverse events during treatment | change from baseline at 3, 6, 9, 12, 18, 24, 30, 36, 42, 48 months and then every 12 months, up to 100 months or if the patient dies, whichever occurs first.
  toxicity will be assessed by the assessment of adverse events related to therapy

SECONDARY OUTCOMES:
hematologic recovery | change from baseline at 3, 6, 9, 12, 18, 24, 30, 36, 42, 48 months and then every 12 months, up to 100 months or until the patient dies, whichever occurs first.
  as measured by complete blood counts
graft failure rate | change from baseline at 3, 6, 9, 12, 18, 24, 30, 36, 42, 48 months and then every 12 months, up to 100 months or until the patient dies, whichever occurs first.
resolution of eosinophilia | change from baseline at 3, 6, 9, 12, 18, 24, 30, 36, 42, 48 months and then every 12 months, up to 100 months or until the patient dies, whichever occurs first.
  as measured by complete blood counts

OTHER OUTCOMES:
regression of antineutrohil cytoplasmic autoantibody (ANCA) titers | change from baseline at 3, 6, 9, 12, 18, 24, 30, 36, 42, 48 months and then every 12 months, up to 100 months or until the patient dies, whichever occurs first.
change in the total lung capacity | change from baseline at 3, 6, 9, 12, 18, 24, 30, 36, 42, 48 months and then every 12 months, up to 100 months or until the patient dies, whichever occurs first.
change in the diffusing capacity of the lungs for carbon monoxide (DLCO) | change from baseline at 3, 6, 9, 12, 18, 24, 30, 36, 42, 48 months and then every 12 months, up to 100 months or until the patient dies, whichever occurs first.
change in the forced expiratory volume (FEV) | change from baseline at 3, 6, 9, 12, 18, 24, 30, 36, 42, 48 months and then every 12 months, up to 100 months or until the patient dies, whichever occurs first.
change in the forced vital capacity (FVC) | change from baseline at 3, 6, 9, 12, 18, 24, 30, 36, 42, 48 months and then every 12 months, up to 100 months or until the patient dies, whichever occurs first.
change in the peak expiratory flow | change from baseline at 3, 6, 9, 12, 18, 24, 30, 36, 42, 48 months and then every 12 months, up to 100 months or until the patient dies, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Mounzer Agha, MD, Principal Investigator — University of Pittsburgh